CLINICAL TRIAL: NCT00716469
Title: Phase I Clinical Study of the Safety of Photodynamic Therapy (PDT) Using Intratumoral Delivery of Non-coherent Light for Photoactivation of LS11 in Children With Plexiform Neurofibromas
Brief Title: Phase I Clinical Study of the Safety of Photodynamic Therapy (PDT) Using LS11 in Children With Plexiform Neurofibromas
Acronym: PDT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is terminated due to expiration of study materials.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Fisher, Assoc. Prof., Children's Hospital of Philadelphia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-10-5008; CHP-856 PDT (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Neurofibroma
Keywords: Neurofibroma; Plexiform; NF1; Photo dynamic therapy
MeSH Terms: conditions — Neurofibroma | interventions — Talaporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LS11 Administration (Experimental): Treatment will be given with a standard 3+3 light dose escalation. The "Treatment Period" will be 28 days. The LS11 dose will be 30mg/m2. The initial light dose will be 50 J/cm. If criteria for dose escalation are met, then the light dose will be escalated to 100J/cm, 150J/cm and 200J/cm. Once the maximum light dose is determined, up to 6 additional patients will be treated at that level to gain further experience with this modality prior to phase II testing. In particular, at least 3 subjects <12 years of age will be enrolled at the maximum tolerable dose (MTD) to allow for further evaluation of safety in younger children. If grade 3 or 4 toxicities are noted at light dose level #1, the LS11 dose will be decreased to 20mg/m2 (2/3 of the standard dose).
  Interventions: Drug: LS11

INTERVENTIONS:
Drug: LS11 — LS11 will be given as a one-time IV infusion over 3-5 minutes.
  Other Names: Talaporfin sodium

SUMMARY:
Plexiform neurofibromas (PN) represent one of the most significant complications of NF1. They are a significant cause of morbidity in neurofibromatosis type 1 (NF1) by causing pain, impaired function, and disfigurement. They may become life-threatening through mechanical compression of vital organs such as the trachea, great vessels, or spinal cord, and may significantly interfere with normal function when located in the extremities or orbit. The only effective therapy for PN is total surgical excision. However, due to local infiltration of normal tissue, gross total resection is usually not feasible, and often PN are completely unresectable due to their location, size, and multiplicity. To date, other therapeutic modalities, including radiotherapy and chemotherapy, have not shown efficacy in PN.

In the present study, local photodynamic therapy will be investigated. Photodynamic therapy (PDT) utilizes a drug, called a photosensitizer or photosensitizing agent, and a particular type of light. When photosensitizers are exposed to a specific wavelength of light, they produce a form of oxygen that kills nearby cells. PDT is expected to result in treatment response with shrinkage of tumor. The main purpose of the study is to determine the maximum amount of light that can be safely used with LS11 for PDT in children with plexiform neurofibromas.

DETAILED DESCRIPTION:
Current treatment options for PN are limited. The only effective therapy for PN is complete surgical resection. Incompletely resected lesions have a high incidence of recurrence, often resulting in the necessity of several surgeries over a patient's lifetime. Development of non-surgical treatments for PN is a high priority. To date, other therapeutic modalities, including radiotherapy and chemotherapy, have not shown efficacy in PN, although it is arguable that these modalities have not been sufficiently studied. Newer approaches, including anti-angiogenesis agents, farnesyl transferase inhibitors, and inhibitors of growth factor pathways are in development and are being studied, but are clearly not proven therapies.

Investigational Agent LS11, talaporfin sodium, was specifically developed as a photosensitizing agent for use in photodynamic therapy. The light activation of LS11 leads to the formation of singlet oxygen causing damage to the vascular endothelial cells leading to vascular thrombosis and occlusion.

Phase I and II studies were conducted in the US and Japan using LS11. PDT with LS11 was generally well tolerated in these studies and there were no serious adverse events noted.

PDT is a novel treatment modality in which a systemically administered photosensitizer (LS11 in our proposal) is activated locally by illuminating the diseased tissue with light of a specific wavelength. Light activation of LS11 leads to the formation of reactive oxygen species that cause damage to the vascular endothelial cells leading to vascular thrombosis and occlusion and subsequently death of tumor cells.

Light Source Placement: Ultrasound may be used to monitor the percutaneous implantation of the Light Source. However, the position of the implanted Light Source must be verified by computed tomography (CT).

* Use a RITA introducer that has a trochar.
* Make a small incision in the skin.
* Insert the introducer into the tumor and advance to the desired position in the target tissue (using ultrasound or CT to verify placement).
* Remove the trochar.
* Insert the Light Source catheter to the end of the sheath. (Avoid mechanical damage to the device, such as twisting, kinking, or exerting force during insertion).
* Pull the sheath back at least 4 centimeters (cm) (the Light Source has to remain in position and not be pulled back with the sheath).
* Verify the Light Source tip location by CT. Reposition if necessary.
* The sheath may be removed completely, after verifying Light Source tip location, at the physician's discretion
* Record distance to lesion surface and to vital structures of the implanted light source.
* Secure the Light Source

LS11 Administration:

* Since compatibility between LS11 and other drugs is not established, LS11 should not be mixed with or physically added to other drugs.
* Every effort should be made to avoid extravasation of LS11 in the surrounding tissue. The extravasated drug may pose prolonged photosensitivity risk to the tissue near the injection site.
* To avoid extravasation, establish an intravenous (IV) line and ensure that there is a free flow of saline or dextrose and water. If a heparin lock is used, flush thoroughly with saline.
* LS11 should be slowly (over 3-5 minutes) administered intravenously as a single dose of 30 mg/m2 or 40 mg/m2.
* Following the injection the line should be flushed with at least 10 cc of saline or dextrose and water.
* In case of extravasation, the site should be thoroughly rinsed with saline or water and carefully bandaged to protect the area from room- and sun-light. The photosensitivity at the extravasated site will last longer than general cutaneous photosensitivity.
* Record the administration start time and end time.

Physical exam, blood tests, electrocardiogram (ECG) and magnetic resonance imaging (MRI) will be performed prior to starting on study and regularly after the treatment per protocol.

Light Exposure Precautions Following PDT-Instructions for Patients: Patients will be sensitive to light and must observe precautions to reduce exposure of skin and eyes to direct sunlight and bright indoor lighting for up to 14 days. The sensitivity to light is due to residual drug that will be present in all parts of the skin and eyes. To minimize skin reactions due to light exposure after LS11 administration, precautions should be taken as detailed in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age: Patients must be ≥ 3 and ≤ 21 years of age.
* Tumor: Patients must have a debilitating, severely disfiguring, life-threatening, or progressive plexiform neurofibroma (PN), which is not surgically resectable and for which there is no other standard medical management.
* Measurable Disease: Patients must have a measurable PN assessed by MRI within 2 weeks prior to starting therapy.
* Tumor Size/Shape/Location:All tumors must:

  1. have a minimum dimension that is ≥ 5 cm in the plane of intended 25mm length Light Source insertion
  2. have a minimum dimension that is ≥ 3.15 cm perpendicular to the plane of intended 25mm length Light Source insertion
  3. be accessible for percutaneous CT (and ultrasound if needed) guided Light Source insertion;
  4. have a shape and location such that the minimum distance between the Light Source and any "critical structure" (defined in section 4.3.4) will be as follows:
* Minimum radial distance = 2.5 cm
* Minimum distance from proximal end of Light Source = 2.5 cm
* Minimum distance from distal end of Light Source = 2 cm
* For patients with NF1: In addition to PN, all study subjects must have at least one other diagnostic criteria for NF1.
* Performance Status: Patients should have a life expectancy of at least 6 months and a Karnofsky (≥ 16 years of age) or Lansky (≤16 years of age) Performance Score ≥ 60.
* Prior/Concurrent Therapy: Patients must have recovered from any specific acute toxicity associated with prior therapy. No concurrent anti-tumor therapy is allowed.
* Laboratory: Patients must have adequate bone marrow, renal, and hepatic function assessed within 7 days prior to start of therapy.

  1. Hematologic:

     Absolute neutrophil count ≥ 1000/ul Platelet count ≥ 100,000/ul Hemoglobin ≥ 8 g/dL PT/PTT ≤ 1.2 times institutional upper limit of normal
  2. Renal: Serum creatinine within upper limit of institutional norm
  3. Hepatic:

Bilirubin ≤ 1.5 times upper limit of normal for age ALT ≤ 2.5 times institutional upper limit of normal for age Albumin ≥ 2 g/dL

* Pregnancy: Female patients of childbearing potential must have negative serum or urine pregnancy test. Patient must not be pregnant or breast-feeding. Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study.
* Informed Consent: All patients or their legal guardians (if the patient is less than 18 years old) must sign an IRB approved document of informed consent indicating their understanding of the investigational nature and the risks of this study before beginning therapy. When appropriate, pediatric patients will be included in all discussions in order to obtain verbal assent.

Exclusion Criteria:

* Patients < 3 or > 21 years of age.
* Tumors that are not debilitating, severely disfiguring, life-threatening, or progressive
* Patients with baseline pain or neuropathy related to their target lesion that is so severe that it effects activities of daily living (i.e. grade 3 or 4).
* Tumors that would require Light Source placement such that a "critical structure" is within the minimum distance required between a "critical structure" and Light Source.
* Tumor that is inaccessible for percutaneous implantation of light source by interventional radiology.
* Patients with a history of porphyria.
* Concomitant use of other drugs known to produce skin photosensitivity (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylureas, thiazide diuretics, and griseofulvin)
* Patients with any serious medical illnesses that, in the investigator's opinion, would compromise a patient's ability to tolerate this therapy.
* Patients receiving any other chemotherapeutics or investigational agents.
* Patients with uncontrolled infections.
* Patients taking NSAIDs or anti-coagulants.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of photodynamic therapy (PDT) for the treatment of plexiform neurofibromas in children. | Week 4 and 12

SECONDARY OUTCOMES:
To evaluate the change in quality of life of treated patients. | Week 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Fisher, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States